CLINICAL TRIAL: NCT02818452
Title: Affecting the Glycemic Impact of Quaker Instant Oatmeal by Adding OatWell28XF: a Dose-Response Study
Brief Title: Glycemic Impact of Oatmeal Plus OatWellXF28
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PEP-1523
Record Dates: First submitted 2016-06-14; First posted 2016-06-29 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Glycemic Responses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Oatmeal containing beta-glucan (Experimental): 27 g oatmeal
  Interventions: Other: Oatmeal
- Oatmeal containing beta-glucan + OatWell28XF Intervention 1 (Experimental): 27.72g oatmeal
  Interventions: Other: Oatmeal + OatWell28XF
- Oatmeal containing beta-glucan + OatWell28XF Intervention 2 (Experimental): 28.43g oatmeal
  Interventions: Other: Oatmeal + OatWell28XF
- Oatmeal containing beta-glucan + OatWell28XF Intervention 3 (Experimental): 29.86g oatmeal
  Interventions: Other: Oatmeal + OatWell28XF
- Oatmeal containing beta-glucan + OatWell28XF Intervention 4 (Experimental): 32.72g oatmeal
  Interventions: Other: Oatmeal + OatWell28XF
- Hot Cereal - Cream of Rice (Placebo Comparator): 20g oatmeal
  Interventions: Other: Hot cereal

INTERVENTIONS:
Other: Oatmeal + OatWell28XF — Intervention involves consumption of one cereal in the beginning of each visit of the crossover sequence
  Arms: Oatmeal containing beta-glucan + OatWell28XF Intervention 1; Oatmeal containing beta-glucan + OatWell28XF Intervention 2; Oatmeal containing beta-glucan + OatWell28XF Intervention 3; Oatmeal containing beta-glucan + OatWell28XF Intervention 4
Other: Oatmeal
  Arms: Oatmeal containing beta-glucan
Other: Hot cereal
  Arms: Hot Cereal - Cream of Rice

SUMMARY:
The objective of this study is to determine the effect on glycemic responses of adding various doses of OatWell28XF to Quaker Instant Oatmeal in order to: 1) describe the dose-response curve and 2) If possible, identify the minimum level of OatWell28XF which, when added to a serving of Quaker Instant Oatmeal, would result in a glycemic response at least 20% less than that elicited by a β-glucan-free cereal.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant females, 18-75 years of age, inclusive
* Body mass index (BMI) ≥ 20.0 and < 35 kg/m² at screening (visit 1).
* Willing to maintain habitual diet, physical activity pattern, and body weight throughout the trial and to refrain from smoking for 12hr prior to each visit.
* Willing to maintain current dietary supplement use throughout the trial. On test days, subject agrees not to take any dietary supplements until dismissal from the GI labs. Failure to comply will result in a rescheduled test visit.
* Normal fasting serum glucose (<7.0mmol/L capillary corresponding to whole blood glucose <6.3mmol/L).
* Willing to abstain from alcohol consumption and avoid vigorous physical activity for 24 h prior to all test visits.
* Absence of health conditions that would prevent fulfillment of study requirements as judged by the Investigator on the basis of medical history.
* Understanding the study procedures and willing to provide informed consent to participate in the study and authorization to release relevant protected health information to the study investigator.

Exclusion Criteria:

* Failure to meet any one of the inclusion criteria
* Known history of AIDS, hepatitis, a history or presence of clinically important endocrine (including Type 1 or Type 2 diabetes mellitus), cardiovascular (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), pulmonary, biliary or GI disorders.
* Use of medications known to influence carbohydrate metabolism, including, but not limited to adrenergic blockers, diuretics, thiazolidinediones, metformin and systemic corticosteroids within 4 weeks of the screening visit, or with any condition which might, in the opinion of Dr. Wolever, the president of GI Testing, either: 1) make participation dangerous to the subject or to others, or 2) affect the results.
* Major trauma or surgical event within 3 months of screening.
* Unwillingness or inability to comply with the experimental procedures and to follow GI Labs safety guidelines.
* Known intolerance, sensitivity or allergy to any ingredients in the study products.
* Extreme dietary habits, as judged by the Investigator (i.e. Atkins diet, very high protein diets, etc).
* Uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg as defined by the average blood pressure measured at screening.
* Change in body weight of >3.5kg within 4 weeks of the screening visit.
* Presence of any signs or symptoms of an active infection within 5 d prior to any test visit. If an infection occurs during the study period, test visits should be rescheduled until all signs and symptoms have resolved and any treatment (i.e. antibiotic therapy) has been completed at least 5 d prior to each test visit.
* History of cancer in the prior two years, except for non-melanoma skin cancer.
* Recent history (within 12 months of screening) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as > 14 drinks per week (1 drink=12 oz beer, 5 oz wine, or 1.5 oz distilled spirits).
* Exposure to any non-registered drug product within 30 d prior to screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Glucose incremental area under the blood glucose response curve | 2 hours post consumption

SECONDARY OUTCOMES:
Peak rise of blood glucose | 2 hours post consumption
Glucose concentrations and increments | 2 hours post consumption
Peak glucose concentration | 2 hours post consumption
Rate of decline of glucose | 2 hours post consumption
Time to return to baseline | 2 hours post consumption

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wolever, MD, Principal Investigator — GI Laboratories
Locations (1):
- GI Labs, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No